CLINICAL TRIAL: NCT04548440
Title: A Phase II Clinical Study of the Efficacy and Safety of Preoperative Sintilimab in Combination With Nab-paclitaxel and Cisplatin in Borderline Resectable Esophageal Squamous Carcinoma
Brief Title: Efficacy and Safety of Preoperative Sintilimab Plus Nab-paclitaxel and Cisplatin in BR-ESCC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry); CSPC Pharmaceutical Group Limited (Industry)
Responsible Party: Principal Investigator, Yuhong Li, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRESCC-Preoperative 02
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — sintilimab; Taxes; Albumin-Bound Paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Sintilimab plus Nab-paclitaxel and Cisplatin (Experimental): Patients receive the following regimen every 3 weeks:
  Sintilimab 200mg IV on Day 1; Albumin-bound paclitaxel 125 mg/m2 IV on Day 1 and Day 8; Cisplatin 75mg/m2 IV on Day 1; Standard hydration regimen on Day 0-3
  After 2-4 cycles, radiological evaluation and multidisciplinary assessment will be performed. If radical resection is possible, surgery is to be performed 3-6 weeks after the last chemotherapy session. In the case of a R0 resection, the investigator will decide whether to perform adjuvant therapy depending on the patient's condition; in the case of R1 or R2 resection, concurrent chemoradiotherapy is recommended. If the multidisciplinary assessment considers that radical resection is not possible, radical concurrent chemoradiotherapy is performed.
  Interventions: Drug: Sintilimab; Drug: Nab paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Sintilimab — Route of administration: Intravenous
  Other Names: Anti-PDCD1 monoclonal antibody IBI308; Tyvyt
Drug: Nab paclitaxel — Route of administration: Intravenously over 30min
  Other Names: Nanoparticle Albumin-Bound Paclitaxel; Abraxane
Drug: Cisplatin — Route of administration: Intravenous
  Other Names: CDDP; Platinol

SUMMARY:
An open-label, non-randomized, phase II study to assess the safety and efficacy of Preoperative Sintilimab Plus Nab-paclitaxel and Cisplatin in Borderline Resectable Esophageal Squamous Cell Carcinoma patients

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the R0 resection rate of Borderline Resectable Esophageal Squamous Cell Carcinoma patients who used preoperative Sintilimab Plus Nab-paclitaxel and Cisplatin

SECONDARY OBJECTIVES:

To evaluate the Pathological Complete Response (pCR) rate, Progression Free Survival (PFS), Relapse Rate, Tumor Regression Grading (TRG) post preoperative chemotherapy, Overall Survival (OS), safety and toxicity of chemotherapy regimen and surgery.

EXPLORATORY OBJECTIVES:

Exploring the benefits of this treatment strategy in Borderline Resectable Esophageal Squamous Cell Carcinoma patients at a molecular level

OUTLINE:

Eligible patients receive Sintilimab and cisplatin intravenously on day 1 and albumin-bound paclitaxel intravenously on days 1 and 8. This cycle is repeated every 3 weeks in the absence of disease progression or unacceptable toxicity. Radiological and multidisciplinary assessment is performed after every 2-4 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide a signed Informed Consent Form
2. Age ≥18 years old
3. Histological confirmation of T4N0-3M0 thoracic esophageal squamous cell carcinoma, absence of distant metastasis and confirmation of a borderline resectable lesion after multidisciplinary assessment using enhanced CT and/or Endoscopic Esophageal Ultrasound or Endobronchial Ultrasound. The definition of a borderline resectable lesion includes: CT showing that the fat gap between the tumor and the aorta is blurred, the angle between three contiguous planes (2mm/layer) and the aorta exceeds 90 degrees; or Endoscopic Esophageal Ultrasound revealing that the tumor has invaded the adventitia layer of the esophagus, and the boundary with the aorta is unclear; or Endobronchial Ultrasound showing an unclear border between the tumor and trachea or bronchus, but has yet invaded the trachea or bronchial mucosa or submucosa
4. Patients have not received any anti-tumor treatment for esophageal cancer (including surgery, chemotherapy, interventional therapy, immunotherapy, radiotherapy, etc.)
5. Life expectancy ≥3 months
6. General physical status (ECOG PS score) 0-1 points
7. Blood routine test (within 7 days): Hb ≥9g/L, NE ≥1.5×109/L, PLT ≥90×109/L
8. Liver and kidney function test (within 7 days): total bilirubin ≤1.5 UNL, creatinine ≤1.5× UNL, AST /ALT ≤2.5xUNL, ALP ≤5.0xUNL
9. No serious complications such as active gastrointestinal bleeding, perforation, jaundice, intestinal obstruction, fever unrelated to malignant disease>38℃
10. Patients with reproductive potential should take effective contraceptive measures
11. Patients with good compliance and that can attend scheduled follow up to assess the efficacy and adverse reactions of the treatment

Exclusion Criteria:

1. Patients with cervical esophageal squamous cell carcinoma
2. Patients with distant metastases
3. Patients with a high risk of complete esophageal obstruction and require interventional therapy
4. Patients with stent implantation in the esophagus or trachea
5. Patients with an esophageal tumor that invaded adjacent organs (aorta or trachea), causing an increased risk of bleeding or perforation, or patients with a fistula
6. Concurrent primary cancers (except for cured skin basal cell carcinoma and cervical carcinoma in situ)
7. History of immunosuppressive drug use within 1 week before treatment, excluding nasal spray, inhalation or use of local glucocorticoids or physiological doses of systemic glucocorticoids (not exceeding 10 mg/day prednisone or equivalent doses of other glucocorticoids) or glucocorticoids used to prevent contrast agent allergy.
8. Patients with active or a past history (within 2 years) of autoimmune disease that need symptomatic treatment (Patient diagnosed with vitiligo, psoriasis, alopecia, or Grave disease that did not require systemic treatment within the past 2 years, hypothyroidism that requires only thyroid hormone replacement therapy and type I diabetes patients treated with insulin replacement therapy only are eligible)
9. Patients with a history of primary immunodeficiency disease
10. Patients with a history of active tuberculosis
11. Patients with a past history of allogenic organ transplantation and allogeneic hematopoietic stem cell transplantation
12. Patients diagnosed with interstitial lung disease that require steroid therapy
13. Patients with a known history of allergy to any monoclonal antibody or chemotherapeutic drugs (taxanes, cisplatin) or their constituents.
14. Patients with a history of severe heart disease, including: history of congestive heart failure, patients with high-risk of uncontrolled arrhythmias, angina pectoris requiring medical treatment, clinically diagnosed heart valve disease, history of severe myocardial infarction and refractory hypertension
15. Patients with chronic diarrhea (4 or more watery stools per day) and patient with renal insufficiency
16. Patients with an active infection or an active infectious disease
17. Neurological or mental disorders that affect cognitive ability
18. Pregnant or breastfeeding women
19. Other acute or chronic diseases, mental diseases or laboratory test values that may cause the following abnormal outcomes: Increase participants or drug administration related risks, interfere with the interpretation of the study results, and patients deemed as ineligible to participate in the study based on the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
R0 resection rate of patients who underwent surgery following preoperative treatment | up to 28 weeks
  The proportion of people with a microscopically margin-negative resection, in which no gross or microscopic tumor remains in the primary tumor bed.

SECONDARY OUTCOMES:
Pathological complete response rate of patients who received surgery following preoperative treatment | up to 28 weeks
  The proportion of patients showing an absence of invasive/in situ cancer after treatment
Progression free survival from the date of first drug administration until the date of first documented progression or date of death, whichever came first. | up to 28 weeks
  The length of time during and after the treatment of the disease, that a patient lives with the disease without its aggravation
Tumor regression rate of patients following preoperative treatment | immediately before surgery
  A decrease in the size of a tumor or the extent of cancer in the body
Relapse rate of patients who received surgery following preoperative treatment | up to 28 weeks
  The number of people with deterioration or recurrence of cancer after a temporary improvement
Overall survival from the date of first drug administration until the date of death from any cause | up to 28 weeks
  The length of time from the start of treatment that patients diagnosed are still alive
Number of patients with adverse events and severity according to NCI CTCAE v5.0 | up to 28 weeks
  Summary of the Adverse events experienced during treatment related to the drug used or surgery in this study

CONTACTS AND LOCATIONS:
Overall Officials: Yuhong Li, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, ICF
Supporting Information: Study Protocol, ICF
Time Frame: When the study complete, the data will become available for 3 years.
Access Criteria: With the permission of professor Yuhong Li